CLINICAL TRIAL: NCT02084940
Title: The Use of a Long Acting GnRH Antagonist (Degarelix) in Controlled Ovarian Hyperstimulation in PCOS Women at a Risk to Developing OHSS Undergoing IVF : a Pilot Study
Brief Title: Long Acting GnRH Antagonist in PCOS Women Undergoing IVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bioroma (Other)
Responsible Party: Sponsor
Other Study IDs: BRM002
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Polycystic Ovarian Syndrome; Ovarian Hyperstimulation Syndrome; Invitro Fertilization
Keywords: PCOS; OHSS; GnRH antagonist; IVF; COH
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GnRH antagonist depot, Degarelix: Women receive 20 mg of Degarelix on the first day of menstrual cycle followed by a fixed dose of 225 IU of recombinant FSH on the second day until the day of ovulation triggering
  Interventions: Drug: GnRH antagonist depot Degarelix

INTERVENTIONS:
Drug: GnRH antagonist depot Degarelix — Women receive 20 mg of Degarelix on the first day of menstrual cycle followed by a fixed dose of 225 IU of recombinant FSH on the second day until the day of ovulation triggering

SUMMARY:
PCOS is a common endocrinopathy affecting 5-10% of women in their reproductive age characterized by hyperandrogenism, chronic anovulation and polycystic ovaries. This syndrome is a serious problem in IVF since there is a high risk of developing ovarian hyperstimulation syndrome (OHSS) during ovarian stimulation with gonadotropins. The introduction of GnRH antagonist in IVF has reduced the incidence of severe OHSS, still maintaining a good ovarian response and pregnancy rate. Recently, a long acting GnRH antagonist, Degarelix, was introduced for prostatic cancer treatment. Furthermore a recent paper reported its use also for the induction of multiple follicular growth in a program of oocyte donation. The aim of this study is to evaluate the feasibility of GnRH antagonist depot use in a protocol of controlled ovarian hyperstimulation in PCOS women at risk of developing OHSS in IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycle (26-39 days)
* primary infertility
* BMI < 30

Exclusion Criteria:

* women with diabetes and other metabolic disease
* women with heart disease
* women with inflammatory or autoimmune disease

Ages: 23 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with PCOS with a previous IVF attempt cancelled due to the risk of OHSS
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | Time Frame: until 12th gestational week
Incidence of OHSS | Time frame: until 7th gestational week

SECONDARY OUTCOMES:
Number of collected oocytes | Time Frame: until 12th gestational week
Estradiol level at HCG day | time frame: until 12th gestational week
Total dose of FSH administered | Time frame: until 12th gestational week
Total days of stimulation | Time frame: until 12th gestational week
implantation rate | time frame: until 12th gestational week

CONTACTS AND LOCATIONS:
Locations (1):
- Bioroma, Rome, Italy, Italy